CLINICAL TRIAL: NCT03934840
Title: A Phase II Study of Carboplatin, Cabazitaxel and Abiraterone in High Volume Metastatic Castration Sensitive Prostate Cancer
Brief Title: CASCARA: Castration Sensitive Carboplatin, Cabazitaxel and Abiraterone
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018LS158; c17-191 (Other: PCCTC)
Record Dates: First submitted 2019-04-26; First posted 2019-05-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; Carboplatin; abiraterone; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carboplatin, Cabazitaxel and Abiraterone (Experimental)
  Interventions: Drug: Cabazitaxel; Drug: Carboplatin; Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: Cabazitaxel — 20 mg/m2 Q 21 days
Drug: Carboplatin — AUC 4 Q21 Days x 6 cycles with ADT
Drug: Abiraterone — 1000 mg PO daily
Drug: Prednisone — 5 mg PO daily on chemotherapy completion

SUMMARY:
This is a phase II clinical trial in patients with metastatic castration sensitive prostate cancer. The objective of the study is to determine the efficacy and further define the safety of the treatment combination. This study will evaluate dose levels of carboplatin AUC 4 with cabazitaxel 20 mg/m2. Patients will be treated with the combination of ADT and carboplatin and cabazitaxel for 6 cycles. After 6 cycles of chemotherapy, they will start abiraterone with ADT. The primary objective is to determine the percent of subjects that have no PSA or radiographic progression at 1 year. Secondary objectives will include determining the progression-free survival, time to PSA nadir and time to PSA progression of carboplatin and cabazitaxel in combination with ADT.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide, or have a legally authorized representative provide, written informed consent and HIPAA authorization for the release of personal health information. A signed informed consent must be obtained before screening procedures are performed.
* Histologically confirmed prostate cancer.
* High volume metastatic disease (defined as the presence of visceral metastases or ≥3 bone lesions).
* ADT for ≤3 months by day 1 of study chemotherapy; Prior episodes of ADT are allowed (i.e. ADT used previously in courses of radiation).
* Testosterone <50 ng/dL. Patients must continue primary ADT with an LHRH analogue if they have not undergone orchiectomy.
* ECOG Performance Status 0 or 1 (see Appendix A)
* Patient has adequate bone marrow and organ function as defined by the following laboratory values:

  * Absolute neutrophil count ≥ 1.5 × 10^9/L
  * Platelets ≥ 100 × 10^9/L
  * Hemoglobin ≥ 9 g/dl
  * Serum creatinine ≤ 1.5mg/dL or estimated creatinine clearance ≥ 50 ml/min
  * In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x ULN. If the patient has liver metastases, ALT and AST <5 x ULN
  * Total bilirubin < ULN; or total bilirubin ≤3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well-documented Gilbert's Syndrome.
* Sexually active males must use a condom during intercourse while taking study drugs and for 30 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid. Fertile males must use a condom with spermicide (double barrier method).
* Age ≥ 18 years

Exclusion Criteria:

* Prior exposure to any chemotherapy, PARPi, or immunotherapy for prostate cancer.
* Prior abiraterone or enzalutamide, unless therapy was for < 2 weeks
* Radiation therapy (including palliative radiotherapy to a metastatic lesion) within 14 days or major surgery (e.g., open abdominal, pelvic, thoracic, orthopedic or neurosurgery) within 28 days of the date of the first dose.
* Other systemic therapies for prostate cancer within 28 days or 5 half-lives, whichever is shorter, prior to day 1 of chemotherapy (with the exception of anti-androgens like bicalutamide).
* PSA <2.0 ng/mL at diagnosis.
* If present, peripheral neuropathy must be ≤ Grade 1
* Patients with an active second malignancy that could, in the investigator's opinion, potentially interfere with the patient's ability to participate and/or complete this trial.
* Patients with central nervous system (CNS) involvement unless they meet ALL of the following criteria:

  * At least 4 weeks from prior therapy completion (including radiation and/or surgery) prior to starting the study treatment
  * Clinically stable CNS tumor at the time of screening.
  * Baseline screening for CNS metastases is not required unless presence of signs and/or symptoms of involvement
* Patients with severe psychiatric illness/social situations that would limit compliance with study requirements in the judgment of treating investigator.
* Patient has a history of non-compliance to medical regimen or inability to grant consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Prostate-Specific Antigen (PSA) or Radiographic Progression | 1 Year
  Proportion of patients who have no PSA or radiographic progression as determined by RECIST 1.1 or PCWG3 criteria

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 1 Year
  Incidence of PFS
PSA Nadir | 1 Year
  Time to time to PSA nadir
Incidence of adverse events | 1 Year
  Safety and Tolerability
Incidence of Homologous Recombination Deficiency (HRD) | 1 Year
  Incidence of HRD
PSA Complete Response Rate | 1 Year
  PSA complete response rate (PSA <0.2 ng/ml) in patient with mutations in DNA repair genes
PSA Complete Response Rate | 1 Year
  PSA complete response rate (PSA <0.2 ng/ml) in patient without mutations in DNA repair genes
PSA Progression | 1 Year
  Time to PSA progression

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Antonarakis, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (8):
- United States (8):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Thomas Jeferson University, Philadelphia, Pennsylvania
  - Lifespan Cancer Institute, Providence, Rhode Island